## **Informed Consent**

I have read this informed consent form.

I had the opportunity to ask questions and all were answered.

I understand that participation in this study is voluntary.

I can choose not to participate in this study, or withdraw after notifying the researcher at any time without being discriminated against or retaliated against, and any of my medical treatment and rights will not be affected as a result.

The study physician may terminate my participation in this study if I require additional treatment, if I do not comply with the study plan, if I suffer a study-related injury, or for any other reason .

I will receive a signed copy of the Informed Consent Form.

| Subject' | s name: |
|-----------|----------------|
| Subject's | signature: |
| date: | year_month day |

I have accurately informed the subject of this document and asked him/her to carefully read this informed consent form and answer the questions or questions raised carefully.

| Researcher' | s name: | <del> </del> |
|----------------|----------------|--------------|
| Investigator's | s signature: | |
| date: | year month day | |

( Note: If the subject is illiterate, a witness signature is required; if the subject is incapacitated, an agent's signature is required )